CLINICAL TRIAL: NCT00214643
Title: A Comparative Assessment of the Efficacy of Fosmidomycin-Clindamycin Versus Sulfadoxine-Pyrimethamine for the Treatment of Children With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Efficacy of Fosmidomycin-Clindamycin for Treating Malaria in Gabonese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Schweitzer Hospital, Netherlands (Unknown)
Collaborators: Albert Schweitzer Hospital (Other)
Organization: Albert Schweitzer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/2005/FOS-CLIN/SP
Record Dates: First submitted 2005-09-11; First posted 2005-09-22 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Malaria
Keywords: Malaria; Fosmidomycin; Clindamycin; Chemotherapy; Gabon
MeSH Terms: conditions — Malaria | interventions — fosmidomycin; Clindamycin

INTERVENTIONS:
Drug: Fosmidomycin — 30 mg/kg
Drug: clindamycin — 10 mg/kg

SUMMARY:
There is a necessity for the development of new malaria drugs. Some antibiotics are also effective against malaria parasites. Fosmidomycin is an antibiotic that has been shown to be effective against malaria, although it cannot achieve a total cure in all patients. Previous small studies have shown that in combination with clindamycin, an commonly used antibiotic, it is highly effective and safe when given for three days, leading to a total cure in most patients. The current study will evaluate its efficacy in a larger population in Gabon, and compare its effect with the generally used drug, sulfadoxine-pyrimethamine.

DETAILED DESCRIPTION:
Fosmidomycin-clindamycin (30 mg/kg and 10 mg/kg) given twice daily for three days is an effective and safe combination of antibiotics which demonstrated good activity against malaria parasite in previous phase II studies in African children. In this phase III trial, the efficacy and safety of the combination will be evaluated in African children with uncomplicated P. falciparum malaria. A single dose of sulfadoxine-pyrimethamine, the standard antimalarial in Gabon, is used as comparator.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated P. falciparum malaria
* P. falciparum asexual parasitaemia between 1,000/µL and 100,000/µL
* Body weight between 10 - 65 kg
* Ability to tolerate oral therapy
* Informed consent, oral assent of the child, if possible
* Residence in study area

Exclusion Criteria:

* Adequate anti-malarial treatment within the previous 7 days
* Antibiotic treatment for the current infection
* Previous participation in this clinical trial
* Haemoglobin < 7 g/dl
* Haematocrit < 23 %
* Leucocyte count > 15,000 /µL
* Mixed plasmodial infection
* Severe malaria (as defined by WHO)
* Any other severe underlying disease (cardiac, renal, hepatic diseases, malnutrition, known HIV infection)
* Concomitant disease masking assessment of response
* History of allergy or intolerance against trial medication

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160
Dates: Start 2005-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Clinical and parasitological cure rate by day 28

SECONDARY OUTCOMES:
Safety and tolerability of the two treatments during the entire study period
Parasite clearance time
Fever clearance time

CONTACTS AND LOCATIONS:
Overall Officials: Saadou Issifou, MD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Background] Kuemmerle HP, Murakawa T, Sakamoto H, Sato N, Konishi T, De Santis F. Fosmidomycin, a new phosphonic acid antibiotic. Part II: 1. Human pharmacokinetics. 2. Preliminary early phase IIa clinical studies. Int J Clin Pharmacol Ther Toxicol. 1985 Oct;23(10):521-8. PMID 4066076
- [Background] Kuemmerle HP, Murakawa T, Soneoka K, Konishi T. Fosmidomycin: a new phosphonic acid antibiotic. Part I: Phase I tolerance studies. Int J Clin Pharmacol Ther Toxicol. 1985 Oct;23(10):515-20. PMID 4066075
- [Background] Rohmer M, Knani M, Simonin P, Sutter B, Sahm H. Isoprenoid biosynthesis in bacteria: a novel pathway for the early steps leading to isopentenyl diphosphate. Biochem J. 1993 Oct 15;295 ( Pt 2)(Pt 2):517-24. doi: 10.1042/bj2950517. PMID 8240251
- [Background] Kuzuyama T, Shizimu T, Takashi S and Seto H. Fosmidomycin, a specific inhibitor of 1-deoxy-D-xylulose 5-phosphate reductoisomerase in the nonmevalonate pathway of isoprenoid biosynthesis. Tetrahaedron Lett 1998;39:7913-6
- [Background] Zeidler J, Schwender J, Müller C, et al. Inhibition of the non-mevalonate 1-deoxy-D-xylulose-5-phosphate pathway of plant isoprenoid biosynthesis by fosmidomycin. Z Naturforsch 1998;53:980-6
- [Background] Lois LM, Campos N, Putra SR, Danielsen K, Rohmer M, Boronat A. Cloning and characterization of a gene from Escherichia coli encoding a transketolase-like enzyme that catalyzes the synthesis of D-1-deoxyxylulose 5-phosphate, a common precursor for isoprenoid, thiamin, and pyridoxol biosynthesis. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2105-10. doi: 10.1073/pnas.95.5.2105. PMID 9482846
- [Background] Takahashi S, Kuzuyama T, Watanabe H, Seto H. A 1-deoxy-D-xylulose 5-phosphate reductoisomerase catalyzing the formation of 2-C-methyl-D-erythritol 4-phosphate in an alternative nonmevalonate pathway for terpenoid biosynthesis. Proc Natl Acad Sci U S A. 1998 Aug 18;95(17):9879-84. doi: 10.1073/pnas.95.17.9879. PMID 9707569
- [Background] Jomaa H, Wiesner J, Sanderbrand S, Altincicek B, Weidemeyer C, Hintz M, Turbachova I, Eberl M, Zeidler J, Lichtenthaler HK, Soldati D, Beck E. Inhibitors of the nonmevalonate pathway of isoprenoid biosynthesis as antimalarial drugs. Science. 1999 Sep 3;285(5433):1573-6. doi: 10.1126/science.285.5433.1573. PMID 10477522
- [Background] Kohler S, Delwiche CF, Denny PW, Tilney LG, Webster P, Wilson RJ, Palmer JD, Roos DS. A plastid of probable green algal origin in Apicomplexan parasites. Science. 1997 Mar 7;275(5305):1485-9. doi: 10.1126/science.275.5305.1485. PMID 9045615
- [Background] Fichera ME, Roos DS. A plastid organelle as a drug target in apicomplexan parasites. Nature. 1997 Nov 27;390(6658):407-9. doi: 10.1038/37132. PMID 9389481
- [Background] Borrmann S, Adegnika AA, Matsiegui PB, Issifou S, Schindler A, Mawili-Mboumba DP, Baranek T, Wiesner J, Jomaa H, Kremsner PG. Fosmidomycin-clindamycin for Plasmodium falciparum Infections in African children. J Infect Dis. 2004 Mar 1;189(5):901-8. doi: 10.1086/381785. Epub 2004 Feb 16. PMID 14976608
- [Background] Borrmann S, Issifou S, Esser G, Adegnika AA, Ramharter M, Matsiegui PB, Oyakhirome S, Mawili-Mboumba DP, Missinou MA, Kun JF, Jomaa H, Kremsner PG. Fosmidomycin-clindamycin for the treatment of Plasmodium falciparum malaria. J Infect Dis. 2004 Nov 1;190(9):1534-40. doi: 10.1086/424603. Epub 2004 Sep 21. PMID 15478056
- [Background] Shulman CE, Dorman EK, Cutts F, Kawuondo K, Bulmer JN, Peshu N, Marsh K. Intermittent sulphadoxine-pyrimethamine to prevent severe anaemia secondary to malaria in pregnancy: a randomised placebo-controlled trial. Lancet. 1999 Feb 20;353(9153):632-6. doi: 10.1016/s0140-6736(98)07318-8. PMID 10030329
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Severe falciparum malaria. World Health Organization, Communicable Diseases Cluster. Trans R Soc Trop Med Hyg. 2000 Apr;94 Suppl 1:S1-90. No abstract available. PMID 11103309
- See also: General information on malaria at the website of the Malaria International Foundation — http://www.malaria.org
- See also: Homepage of the Medical Research Unit, Lambaréné — http://www.lambarene.org